CLINICAL TRIAL: NCT00417586
Title: New Ultrasound Instrument for Carotid Screening
Brief Title: Cost-Effectiveness of a Specialized Ultrasound Instrument to Diagnose Carotid Stenosis as a Way to Reduce the Risk of Stroke
Status: Completed | Type: Observational
Sponsor: DVX, LLC (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Vilkomerson, President, DVX, LLC
Other Study IDs: 468; R44HL072534 (NIH); R44HL072534-02A1 (NIH)
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Carotid Stenosis; Cerebrovascular Accident
Keywords: Stroke
MeSH Terms: conditions — Carotid Stenosis; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Specialized Doppler Ultrasound Instrument — Patients with a reading of 140 cm/sec or higher will be referred for further duplex screening

SUMMARY:
Carotid stenosis, a condition in which plaque builds up inside the arteries of the neck and blocks blood flow to the brain, is one common cause of stroke. This study will evaluate the cost-effectiveness of using a new, specialized ultrasound device to screen individuals who are at risk for carotid stenosis.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death, and the leading cause of long-term disability in the United States. At least half of all strokes are caused by carotid stenosis, a condition in which the arteries in the neck become blocked with plaque and harden. Plaque that breaks off the carotid artery wall and travels to the brain can block critical blood vessels, possibly resulting in a stroke. Carotid endarterectomy, a procedure that removes plaque buildup, can greatly reduce an individual's risk for stroke. Currently, the conventional duplex Doppler ultrasound examination that is used to screen for carotid stenosis requires a skilled sonographer or physician, and is therefore expensive. Study researchers have developed a more cost-effective option: a specialized ultrasound instrument specifically designed to perform carotid stenosis screenings and meant to be used by non-specialist nurses. Previous research has shown that this instrument is inexpensive, easy to use, and effective at diagnosing carotid stenosis. The purpose of this study is to evaluate the cost-effectiveness of the alternative ultrasound instrument at screening older adults who are at risk for carotid stenosis. If the instrument is shown to be cost-effective, it may eventually lead to widespread screening and a reduced incidence of stroke.

In this study, nurses in selected physician's offices will be trained to use the carotid ultrasound screening instrument. Patients over 65 years of age with at least one risk factor for carotid stenosis but with no symptoms will be screened with the device. Screening will take place in the doctors' offices or, when more convenient, at a central screening location; however, in all cases the nurses will use the instrument rather than specialized ultrasound technologists. Individuals found to have carotid stenosis will be referred to undergo a conventional duplex Doppler ultrasound examination for a definitive diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* At least one risk factor for carotid stenosis (e.g., cardiac disease, elevated cholesterol, smoking, hypertension)

Exclusion Criteria:

* Any symptoms or indications of carotid stenosis or stroke

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Primary care patients who fit inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 984 (Actual)
Dates: Start 2007-06; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Goldman, MD, Principal Investigator — Princeton Surgical Associates
Locations (1):
- Princeton Surgical Associates, Princeton, New Jersey, United States